CLINICAL TRIAL: NCT04591366
Title: Barrier-Protect Study: Do Barrier Dressings Reduce Device Infection: a Pilot, Randomized Controlled Trial
Brief Title: Barrier-Protect Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20200369-01H
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Infection
Keywords: Cardiac; Device
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants and staff taking the swab will be blinded as to the randomization allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard skin prep prior to procedure will be performed and an adhesive iodine-infused barrier dressing will be applied post procedure but prior to taking the culture swab and closing the incision.
  Interventions: Other: Barrier dressing
- Intervention (Experimental): Standard skin prep prior to procedure plus an adhesive iodine-infused barrier dressing prior to incision, post procedure a culture swab will be taken and the incision closed.
  Interventions: Other: Barrier dressing

INTERVENTIONS:
Other: Barrier dressing — A barrier dressing will be applied either pre or post implant prior to a culture swab and closing the incision.

SUMMARY:
This study will evaluate the effect of an iodine impregnated barrier dressing on device pocket swab culture positivity. Minimizing contamination during the implant procedure can be one of the potential improvements to prevent CIED infections. Patients requiring a lead change, battery change or device upgrade will be eligible. This is a randomized, blinded study where participants will be randomized to having the barrier dressing applied before any incision is made (experimental group) or applying the dressing just prior to collecting the culture swab (control group). Patients and the staff taking the culture swab at the end of the procedure are blinded as to which group the participant is randomized to.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18
2. Second or later procedure (including pulse generator change, lead revision and device upgrade procedures) involving manipulation of the pre-existing device pocket.
3. PADIT risk score ≥ 5

Exclusion Criteria:

1. Unable or unwilling to provide informed consent.
2. De novo device implantation.
3. Active device infection.
4. Iodine allergy
5. Life expectancy less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
End of surgery pocket swab culture positivity | one month post procedure
  To investigate end of procedure pocket swab culture positivity as a potential surrogate marker of device infection

SECONDARY OUTCOMES:
CIED infection, defined as in the recent PADIT trial | Year 1 and 2 post procedure
  1. Pocket infection: Nosocomial surgical site infection will be defined according to the 2008 National Healthcare Safety Network (NHSN) and US CDC definitions for superficial and deep surgical site infections (30)
  2. Endocarditis will be diagnosed according to the Modified Dukes' criteria (31). These were adapted by Klug D et al. to diagnose endocarditis in patients with implantable cardiac devices (32).
  3. Bloodstream infections will be defined according to 2008 NHSN and US CDC definitions for Primary bloodstream infections (33)

CONTACTS AND LOCATIONS:
Overall Officials: Alper Aydin, Dr., Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aydin A, Golian M, Klein A, Redpath C, Davis DR, Ramirez FD, Nair GM, Green MS, Sadek M, Nery PB, Hansom SP, Al Hinai G, Weng W, Berbenetz N, Thibert MJ, Salmeen Y, Martow E, Tan LW, Almidani G, Alshehri A, Alzahrani A, Alharbi F, Corrales-Medina V, Wells GA, Birnie DH. Iodinated Adhesive Drapes for Repeat Cardiac Implantable Device Implantation: A Randomized Clinical Trial. JAMA Cardiol. 2025 Oct 1;10(10):1016-1023. doi: 10.1001/jamacardio.2025.2835. PMID 40864462